CLINICAL TRIAL: NCT06640049
Title: A Phase 2, Single-Arm, Open-Label Study With Dostarlimab Monotherapy in Participants With Untreated Stage II/III dMMR/MSI-H Locally Advanced Rectal Cancer in China
Brief Title: A Study of Dostarlimab in Participants With Untreated Locally Advanced Rectal Cancer in China
Acronym: China AZUR-1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 221972
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Neoplasms, Rectal
Keywords: Dostarlimab; GSK4057190A; TSR-042; Rectal cancer; dMMR; MSI-H
MeSH Terms: conditions — Rectal Neoplasms | interventions — dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dostarlimab monotherapy (Experimental): Participants will receive dostarlimab as monotherapy.
  Interventions: Biological: Dostarlimab

INTERVENTIONS:
Biological: Dostarlimab — Dostarlimab will be administered.
  Other Names: GSK4057190A; TSR-042

SUMMARY:
The main goal of this study is to evaluate the effect of dostarlimab monotherapy in Chinese participants with locally advanced Mismatch-repair deficient (dMMR)/ Microsatellite instability-high (MSI-H) rectal cancer who have received no prior treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participant has histologically confirmed Stage II to III (T3-T4, N0, or T any, N+), locally advanced rectal adenocarcinoma
* Participant has radiologically and endoscopically evaluable disease
* Participant has a tumor which can be categorized as dMMR or MSI-H by central assessment

Exclusion Criteria:

* Participant has distant metastatic disease
* Participant has received prior radiation therapy, systemic therapy, or surgery for management of rectal cancer
* Has a known additional malignancy that progressed or required active treatment within the past 2 years
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* Has experienced any of the following with prior immunotherapy: any irAE ≥ Grade 3, immune-related severe neurologic events of any-grade (e.g., myasthenic syndrome/myasthenia gravis, encephalitis, Guillain Barré Syndrome, or transverse myelitis), exfoliative dermatitis of any grade [SJS (Stevens-Johnson Syndrome, TEN (Toxic Epidermal Necrolysis), DRESS (Drug rash with eosinophilia and systemic symptoms)], or myocarditis of any grade. Non-clinically significant laboratory abnormalities are not exclusionary
* Has any history of interstitial lung disease or pneumonitis
* Has received or plans to receive an organ or stem cell transplant that uses donor stem cells (allogeneic stem cell transplant)
* Has a history of severe allergic and/or anaphylactic reactions to chimeric, human, or humanized antibodies, fusion proteins, or known allergies to dostarlimab, or its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-10-17 (Actual); Primary Completion 2027-10-24 (Estimated); Study Completion 2031-04-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Sustained Complete Clinical Response for 12 Months (cCR12) as assessed by Independent Central Review (ICR) | 18 months
  cCR12 is achieved when a participant maintains complete clinical response (cCR) as assessed by Independent central review (ICR) for 12 months from the first disease assessment after last dose of study intervention. Timeframe calculation includes 6 months (9 cycles of dostarlimab, with each cycle lasting 21 days) plus an additional 12 months of assessment time, amounting to a total of 18 months.

SECONDARY OUTCOMES:
Number of Participants with Sustained Complete Clinical Response for 24 Months (cCR24) as assessed by ICR | 30 months
  cCR24 is achieved when a participant maintains cCR as assessed by ICR for 24 months following their first disease assessment after last dose of study intervention. Timeframe calculation includes 6 months (9 cycles of dostarlimab, with each cycle lasting 21 days) plus an additional 24 months of assessment time, amounting to a total of 30 months.
Number of Participants with Sustained Complete Clinical Response for 36 Months (cCR36) as assessed by ICR | 42 months
  cCR36 is achieved when a participant maintains cCR as assessed by ICR for 36 months following first disease assessment after last dose of study intervention. Timeframe calculation includes 6 months (9 cycles of dostarlimab, with each cycle lasting 21 days) plus an additional 36 months of assessment time, amounting to a total of 42 months.
Number of Participants with Event Free Survival at 3 years (EFS3) as assessed by Investigator | 3 years
  EFS3 is defined as participants who remained alive and free of disease progression precluding surgery, local recurrence, and distant recurrence at 3 years from the first dose of study intervention as assessed by Investigator.
Event Free Survival (EFS) as assessed by Investigator | Up to approximately 77 months
  EFS is defined as time from the date of first dose of study intervention to any of the following events including progression of disease that precludes surgery, local recurrence, distant recurrence (all as assessed by the investigator), or death due to any cause.
Number of Participants with cCR12 as assessed by Investigator | 18 Months
  cCR12 is achieved when a participant maintains cCR as assessed by Investigator for 12 months from the first disease assessment after last dose of study intervention. Timeframe calculation includes 6 months (9 cycles of dostarlimab, with each cycle lasting 21 days) plus an additional 12 months of assessment time, amounting to a total of 18 months.
Number of Participants with cCR24 as assessed by Investigator | 30 Months
  cCR24 is achieved when a participant maintains cCR as assessed by Investigator for 24 months from the first disease assessment after last dose of study intervention. Timeframe calculation includes includes 6 months (9 cycles of dostarlimab, with each cycle lasting 21 days) plus an additional 24 months of assessment time, amounting to a total of 30 months.
Number of Participants with cCR36 as assessed by Investigator | 42 Months
  cCR36 is achieved when a participant maintains cCR as assessed by Investigator for 36 months from the first disease assessment after last dose of study intervention. Timeframe calculation includes 6 months (9 cycles of dostarlimab, with each cycle lasting 21 days) plus an additional 36 months of assessment time, amounting to a total of 42 months.
Objective Response Rate (ORR) assessed by ICR | Up to 37 Weeks
  ORR is defined as number of participants achieving a partial response (PR), near complete response (nCR) or cCR at post-intervention disease assessment (PIDA) or at least 4 weeks but no longer than 8 weeks after PIDA for participants with nCR or incomplete clinical response (iCR) (PIDA 2) as assessed by ICR.
Objective Response Rate (ORR) as assessed by Investigator | Up to 37 Weeks
  ORR by Investigator is defined as number of participants achieving a PR, nCR, or cCR at PIDA.
Organ Preservation Rate | Up to 3 years
  Organ Preservation Rate is defined as number of participants who did not undergo any rectal cancer surgery either as primary management or for local recurrence, or who did not have a permanent colostomy created, at any time up to 3 years.
Disease-Specific Survival (DSS) | Up to approximately 77 months
  DSS is defined as time from the date of first dose of study intervention to death due to disease under study.
Disease-Specific Response at 5 years (DSS5) | Up to 5 years
  DSS5 is defined as the number of participants not dying due to disease under study at 5 years from the first dose of study intervention.
Overall Survival (OS) | Up to approximately 77 months
  OS is defined as time from first dose of study intervention to death from any cause.
Overall Survival at 5 years (OS5) | Up to 5 years
  OS5 is defined as number of participants being alive at 5 years from first dose of study intervention.
Number of Participants with Adverse Events (AEs), Serious Adverse Events (SAEs), Immune related Adverse Events (irAEs) and AEs leading to death or discontinuation of study intervention. | Up to approximately 77 months
Serum concentration of Dostarlimab | Up to approximately 77 months
Concentration at the end of infusion (C-EOI) of Dostarlimab | Up to approximately 77 months
Trough Concentration (C-trough) of Dostarlimab | Up to approximately 77 months
Number of Participants with Anti-Drug Antibodies (ADA) against Dostarlimab | Up to approximately 77 months

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - GSK Investigational Site, Chengdu
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Jinan
  - GSK Investigational Site, Kunming
  - GSK Investigational Site, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/